CLINICAL TRIAL: NCT00629473
Title: A Phase 1 Clinical Trial of NPI-0052 in Patients With Advanced Malignancies
Brief Title: Phase 1 Clinical Trial of NPI-0052 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI-0052-102
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Advanced Cancer
Keywords: multiple myeloma; leukemias (inc. CLL); lymphomas; cutaneous lymphoma; marginal zone lymphoma; advanced malignancies without standard treatment options
MeSH Terms: conditions — Multiple Myeloma; Leukemia; Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone | interventions — marizomib; Proteasome Inhibitors; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm AM: advanced malignancies (Experimental): Dose Escalation - 9 dose cohorts NPI-0052 on Days 1, 8, 15 every 28 days NPI-0052 doses ranging from 0.1 to 0.9 mg/m2
  Interventions: Drug: NPI-0052 on Days 1, 8, 15 every 28 days
- Arm MM: multiple myeloma (Experimental): Dose Escalation - 8 dose cohorts NPI-0052 on Days 1, 4, 8, 11 every 21 days NPI-0052 doses ranging from 0.075 to 0.6 mg/m2 Dexamethasone 20 mg oral or IV day before and day after NPI-0052 dosing.
  Interventions: Drug: NPI-0052 on Days 1, 4, 8, 11 every 21 days; Drug: Dexamethasone

INTERVENTIONS:
Drug: NPI-0052 on Days 1, 8, 15 every 28 days — NPI-0052 dose ranging from 0.1 to 0.9 mg/m2 NPI-0052 IV injection over 1 to 120 minutes on Days 1, 8, and 15 of 4-week cycles
  Other Names: marizomib; proteasome inhibitor
  Arms: Arm AM: advanced malignancies
Drug: NPI-0052 on Days 1, 4, 8, 11 every 21 days — NPI-0052 dose ranging from 0.075 to 0.6 mg/m2 NPI-0052 IV injection over 1 to 120 minutes on Days 1, 4, 8, and 11 of 3-week cycles
  Other Names: marizomib; proteasome inhibitor
  Arms: Arm MM: multiple myeloma
Drug: Dexamethasone — 20 mg oral or IV day before and day after NPI-0052 dosing.
  Other Names: Decadron
  Arms: Arm MM: multiple myeloma

SUMMARY:
This is a Phase 1 clinical trial examining the safety, pharmacokinetics and pharmacodynamics of escalating doses of the proteasome inhibitor NPI-0052 in patients with advanced malignancies including solid tumors, lymphomas, leukemias and multiple myeloma. By inhibiting proteasomes NPI-0052 prevents the breakdown of proteins involved in signal transduction, which blocks growth and survival in cancer cells.

DETAILED DESCRIPTION:
Patients were enrolled in 1 of 2 study arms. Arm AM (weekly doses of NPI-0052) consisted of patients with solid and hematological malignancies excluding multiple myeloma (MM), and these patients received NPI-0051 once weekly for 3 weeks of every 4 weeks. Arm MM (twice-weekly doses of NPI-0052) consisted of patients with MM and other hematological malignancies, and these patients received NPI-0052 twice weekly for 2 weeks of every 3 weeks. All patients received NPI-0052 administered IV over approximately 1 to 120 minutes. Patients with MM (Arm MM) also received 20 mg dexamethasone per orally or IV on the day before and the day of NPI-0052 dosing.

Patients were initially enrolled in dose-escalating cohorts to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of NPI-0052. Once the RP2D was determined for each arm of the study, the RP2D was evaluated in the dose-expansion stage of the study.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Status (KPS) > 70%.
* Histologically-confirmed advanced malignancy for which a standard, approved therapy is not available.
* Adequate renal, liver, pancreatic and hematologic function
* Signed informed consent (sample IC form is provided in Appendix A).

Exclusion Criteria

* Administration of chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic) within 28 days
* Patients that require G-CSF and/or platelet support during screening and are likely to require G-CSF and/or platelet support for the duration of the clinical trial.
* Patients with ongoing coagulopathies and/or taking anticoagulants
* Patients receiving intrathecal therapy.
* Known brain metastases.
* Pre-existing adrenal insufficiency; concomitant therapy with replacement corticosteroids. Pre-existing acute or chronic pancreatitis.
* Significant cardiac disease.
* Pregnant or breast-feeding women.
* Concurrent, active secondary malignancy for which the patient is receiving therapy. (Lymphoma patients with a diagnosis of a potentially hormone-sensitive tumor who are without evidence of disease for this second malignancy may continue to receive hormonal therapy).
* Patients with proteinuria Grade 2 or greater
* Active uncontrolled bacterial or fungal infection requiring systemic therapy; infection requiring parenteral antibiotics.
* Patients who are known to be HIV positive or have active Hepatitis A, B, or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of NPI-0052 | Cycle 1 (Arm AM: 28-days, Arm MM: 21-days)
  Assess dose-limiting toxicities during Cycle 1 for each treatment arm

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics activity of NPI-0052 | Baseline, Days 1 and 15 (before injection and 1 hour post injection) of Cycle 1
  the assess the time course of NPI-0052 in the body
To evaluate the safety and tolerability of NPI-0052 | Treatment period through 28-days after the last dose of study drug
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
To evaluate the pharmacodynamics of NPI-0052 | Baseline, Days 1 and 15 (before injection and 1 hour post injection) of Cycles 1 and 2 and of every other cycle thereafter through study completion
  proteasome inhibition in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Reich, MD, Study Director — Triphase Research and Development I Corp
Locations (7):
- Australia (7):
  - Mater Adult Hospital, South Brisbane, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancen Center, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital and University of Western Australia, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided